CLINICAL TRIAL: NCT06828536
Title: Female Genital Schistosomiasis in Migrant Women: A Pilot Study
Acronym: GynoBizh
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP240729
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Diagnostic; Schistosomiasis
Keywords: femal genital schistosomiasis; migrant women; colposcopy; Diagnostic pilot study; Schistosoma spp. PCR
MeSH Terms: conditions — Disease; Schistosomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group (Experimental)
  Interventions: Other: Gynecology consultation; Other: Transvaginal ultrasound; Other: PCR Schistosoma spp

INTERVENTIONS:
Other: Gynecology consultation — Gynecology consultation M0 - M3 - M6 - M12
Other: Transvaginal ultrasound — Transvaginal ultrasound
Other: PCR Schistosoma spp — PCR Schistosoma spp Colposcopy Cervical biopsy Cervical smear

SUMMARY:
This pilot study, "GynoBizh," investigates the frequency and clinical characteristics of female genital schistosomiasis (FGS) among migrant women from sub-Saharan Africa living in non-endemic countries. Schistosomiasis is a significant global parasitic disease, with a high seroprevalence in migrants. The study aims to assess the presence of genital lesions through gynecological examinations, colposcopy, and molecular tests, identifying diagnostic markers and associated health conditions. Fifty participants will be followed over a year to improve understanding and management of FGS in underserved populations.

DETAILED DESCRIPTION:
Female genital schistosomiasis (FGS) is an underdiagnosed and under-researched condition, particularly in non-endemic regions, despite its significant prevalence among migrant women from sub-Saharan Africa. Schistosomiasis is the second most common parasitic disease globally, with a seroprevalence of up to 25% among migrants from endemic regions. FGS, characterized by genital lesions, often goes unrecognized due to a lack of awareness among healthcare providers in non-endemic countries and the absence of a gold-standard diagnostic method.

This pilot study, conducted at Bicêtre Hospital by Assistance Publique - Hôpitaux de Paris, seeks to evaluate the frequency of FGS-related genital lesions in a cohort of 50 women aged 25-65 years. Participants, all seropositive for schistosomiasis and originating from sub-Saharan Africa, will be recruited over six months and followed for one year. The study involves a comprehensive diagnostic approach, including gynecological examinations, colposcopy, endovaginal ultrasounds, and molecular tests (e.g., PCR on vaginal self-samples and cervical smears). Lesions identified during initial exams will be reassessed at follow-ups scheduled at 3, 6, and 12 months.

Secondary objectives include documenting participants' gynecological and obstetric histories, symptoms, and potential co-infections with HIV, HBV, and HCV. The study will also compare the effectiveness of different diagnostic tools for FGS and explore the presence of Schistosoma DNA in plasma and genital samples. Data will be collected through clinical assessments, questionnaires, and laboratory analyses, with results analyzed using robust statistical methods.

While the procedures are minimally invasive, risks are low and limited to mild discomfort from colposcopy and minor bleeding following biopsies. This study is expected to yield valuable insights into the prevalence and characteristics of FGS in non-endemic settings, addressing an overlooked health issue that disproportionately affects migrant women. By highlighting diagnostic challenges and identifying effective tools, this research aims to inform clinical guidelines, improve care, and advocate for targeted public health strategies for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 to 65 years
* Born in a schistosomiasis-endemic area in sub-Saharan Africa
* With a positive serology by Schistosoma spp. Western Blot

Exclusion Criteria:

* Refusal to participate in the study
* Patient unable to provide consent
* Patient under guardianship or trusteeship
* Patient who is a virgin at the time of selection
* Patient who is pregnant at the time of selection

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
To determine the frequency of lower genital involvement due to schistosomiasis (perineum, vulva, vagina, cervix) in women born in endemic areas in sub-Saharan Africa and living in non-endemic countries who have positive serology for schistosomiasis | 12 months
  The frequency of lower genital involvement in women who are seropositive for schistosomiasis, as seen on gynaecological examination of the vulva, vagina and cervix using the speculum and of the cervix using colposcopy, carried out during the dedicated gynaecology consultation prior to treatment

SECONDARY OUTCOMES:
Take a gynaecological history of schistosomiasis-positive women with or without proven FGS (gestational age, parity, miscarriages, ectopic pregnancies, infertility, HPV infection, upper genital infection) | inclusion
  Personal gynaecological history: number of pregnancies, number of children, miscarriages, ectopic pregnancies, percentage of infertility (defined as no pregnancy after 1 year of the trial), number of HPV infections (condyloma, cervical dysplasia), number of upper genital infections, etc.
Describe the gynaecological and urological symptoms of patients infected with schistosomiasis | inclusion
  Percentage of women with urological symptoms: dysuria, burning, nocturia, pollakiuria, macroscopic haematuria, microscopic haematuria
Describe the specific clinical lesions of FGS on colposcopy and vulvar and endovaginal examination | inclusion
  Percentage of women with gynaecological symptoms: vulvar pruritus, abnormal leucorrhoea, menometrorrhagia, dyspareunia, dysmenorrhoea, pelvic pain, etc.
To describe the ultrasound lesions of the genital tract found in patients who are seropositive for schistosomiasis | inclusion
  Percentage of women with ultrasound genital tract lesions compatible with schistosomiasis
Compare positivity rates of tests for FGS: (i) Schistosoma spp. PCR on vaginal self-sampling, (ii) lesions at colposcopy, (iii) Schistosoma spp. PCR on cervical/vaginal smears, (iv) cervical biopsy, (v) egg detection on cervical/vaginal smears | inclusion
  Percentage of women with a positive test among : (i) Schistosoma spp. PCR on vaginal self-sampling, (ii) specific lesions seen at colposcopy, (iii) Schistosoma spp. PCR on cervical and vaginal smears, (iv) cervical biopsy, (v) egg testing on cervical and vaginal smears
Determining the presence of HIV, HBV and HCV co-infection | inclusion
  Percentage of co-infection by determination of HIV, HBV, HCV serology
To determine the presence of Schistosoma spp. DNA in plasma in the event of positive serology in this context of chronic bilharzian infection | inclusion
  Percentage of positive Schistosoma spp PCRs on vaginal self-sampling and Number of patients with Schistosoma spp PCR in serum

IPD SHARING:
Plan to Share IPD: No